CLINICAL TRIAL: NCT01150214
Title: DECAAF: DE-MRI Determinant of Successful Radiofrequency Catheter Ablation of Atrial Fibrillation
Brief Title: DECAAF: Delayed-Enhancement MRI (DE-MRI) Determinant of Successful Radiofrequency Catheter Ablation of Atrial Fibrillation
Acronym: DECAAF
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Nassir F. Marrouche, MD, Associate Professor, University of Utah
Other Study IDs: IRB_00039522
Record Dates: First submitted 2010-06-22; First posted 2010-06-24 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; af; magnetic resonance imaging; mri; left atrium; fibrosis; structural remodeling
MeSH Terms: conditions — Atrial Fibrillation; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- DE-MRI: All patients will undergo Delayed-Enhancement Magnetic Resonance Imaging (DE-MRI)to quantify the degree of atrial structural remodeling or fibrosis pre-ablation and DE-MRI will be obtained at 3, 6, and 12 months follow-up to detect and quantify ablation-related scar formation.
  Interventions: Procedure: DE-MRI

INTERVENTIONS:
Procedure: DE-MRI — Using Delayed-Enhancement Magnetic Resonance Imaging (DE-MRI) to identify fibrotic and scarred cardiac tissue. DE-MRI is a non-invasive method of identifying the extent and the distribution of structural remodeling or fibrosis and scarring associated with atrial fibrillation both pre- and post-ablation.

SUMMARY:
This is a multi-center, observational, 1-year prospective cohort study (1 year follow-up, at 3, 6 and 12 month) with approximately 675 participants. We will conduct a thorough outcomes assessment utilizing data from Magnetic Resonance Imaging (MRI) scans, as well as pre-procedure and follow-up data. Scans will be blinded to location of participating site. MRI scans will be sequenced and analyzed as they arrive from the database.

Imaging Protocol: All patients will undergo a Delayed-Enhancement MRI (DE-MRI) within 30 days prior to the atrial fibrillation (AF) ablation procedure. The purpose of the initial MRI is to quantify the degree of atrial structural remodeling or fibrosis pre-ablation. Following ablation, DE-MRI will be obtained at 3, 6, and 12 months follow-up to detect and quantify ablation-related scar formation.

Clinical Follow-up: The institution where the ablation was performed will continue post-procedural care following standard of care procedures.

Atrial arrhythmia recurrences will be catalogued up to one year post-ablation and predictors of recurrences of AF will be determined by statistical analysis. The specific mechanism and electrophysiological characteristics of atrial arrhythmia recurrence will also be analyzed.

Our hypotheses are (1) DE-MRI will reproducibly stage the progression left atrium fibrosis in AF; (2) DE-MRI will reproducibly aid in quantifying and identifying the distribution of catheter ablation-related scarring in the left atrium; and (3) the stage of left atrium fibrosis pre-ablation and the amount and location of scarring will predict success of catheter ablation therapy for AF.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is an electrophysiological condition characterized by a disorganized electrical activity in the atria of the heart. AF is associated with structural heart disease including hypertension, systolic and diastolic ventricular dysfunction and valvular heart disease. It represents a significant public health problem with the increasing longevity of the general population. A major determinant of the progression of AF is structural remodeling or fibrosis that occurs in the left atrium. A more extensively remodeled atrium represents the substrate needed for the arrhythmia to persist. Structural remodeling is also a major determinant for success of rhythm control strategies in AF. While catheter ablation has been reproducibly shown to be superior to anti-arrhythmic drug therapy for rhythm control in AF, the success of this procedure is significantly affected by the extent of structural remodeling present at the time of catheter ablation.

Delayed-Enhancement Magnetic Resonance Imaging (DE-MRI) has been demonstrated to be a very effective modality in identifying fibrotic and scarred cardiac tissue with excellent correlation with autopsy findings. This is related to the characteristics of Gadolinium, an extracellular contrast agent that is very effective in identifying regions of fibrotic non-viable myocardium. DE-MRI technology can be a very powerful, non-invasive method, of identifying the extent and the distribution of structural remodeling or fibrosis associated with AF.

Applying DE-MRI technology to the atrium causes significant technical challenges. The atrial wall is often a few millimeters thick which requires high spatial resolution to obtain adequate and useful images. In addition, image acquisition has to be gated to the diastolic phase of the atrial contraction cycle, which may be difficult to do when the patient is in AF. The ongoing research at the University of Utah has shown significant progress and very promising results overcoming the challenges mentioned. Specific image acquisition sequences have allowed for reproducible identification of high pixel intensity regions within the 2-dimensional images of the atrial wall. Three-dimensional reconstruction of the entire left atrium then provides a quantification of the overall volume occupied by these hyper-enhanced regions relative to the entire left atrial wall volume. Used prior to catheter ablation, DE-MRI can therefore identify regions of significant structural remodeling or fibrosis. The same technology has also been shown to be very useful in examining the amount and distribution of ablation related scarring.

Clinical patient characteristics will be collected for this study from clinic visits and chart reviews.

Imaging Protocol: All patients will undergo a DE-MRI within 30 days prior to the AF ablation procedure using a DE-MRI protocol. The purpose of the initial MRI is to quantify the degree of atrial structural remodeling or fibrosis pre-ablation. Following ablation, DE-MRI will be obtained at 3, 6, and 12 months follow-up to detect and quantify ablation-related scar formation (Figs. 4-5).

Clinical Follow-up: The institution where the ablation was performed will continue post-procedural care following standard of care procedures. Monitoring and definition of atrial arrhythmia AF recurrences will be guided by the HRS consensus document on ablation of atrial fibrillation.

Clinical and MRI data will be stored using the IRB-approved University of Utah database. De-identified clinical data and MRI images from participating institutions will also be submitted to the database, and will be processed at the University of Utah for pre- and post-ablation fibrosis and scar quantification. The ablation strategy utilized and procedural endpoint will be left to the discretion of the operators at the participating sites. This data will also be collected and included in the final analysis. MRI image processors at the University of Utah will be blinded to the ablation technique and mother institution using a unique de-identified study participant ID number.

Atrial arrhythmia recurrences will be catalogued up to one year post-ablation and predictors of recurrences determined by multivariate/survival analysis. The specific mechanism and electrophysiological characteristics of atrial arrhythmia recurrence will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent an AF ablation as per recent Heart Rhythm Society (HRS) consensus document, as per the University of Utah AFIB Database (IRB_00020347)
* Patients who have had an MRI post-ablation.
* Age ≥18 years.

Exclusion Criteria:

* Contraindication for DE-MRI with a full dose of Gadolinium-based contrast agent.
* Previous left atrial ablation or surgical procedure
* Renal failure with CrCl <60 ml/min
* Women currently pregnant, breastfeeding, or of childbearing age not currently taking or not willing to use a reliable form of contraception
* Mental or physical inability to take part in the study
* Uncontrolled hypertension
* Morbid obesity (BMI > 35), or inability to be placed in MRI due to body mass.
* Patients who have not had a DE-MRI post-ablation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of those patients who have undergone catheter ablation for atrial fibrillation.
Sampling Method: Non-Probability Sample
Enrollment: 339 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Relationship between extent of pre-ablation fibrosis and recurrence post-ablation | 1 year
  The percentage of pre-ablation fibrosis in atrial fibrillation patients can significantly impact the incidence of recurrences post-ablation.

SECONDARY OUTCOMES:
Relationship between extent of Post-ablation scar and incidence of atrial fibrillation recurrences post-catheter ablation for AF | Post-ablation scar
  The extent of lesions created by ablation may have an impact on the incidence of recurrence of AF post-ablation

CONTACTS AND LOCATIONS:
Overall Officials: Nassir F Marrouce, MD, FHRS, Principal Investigator — CARMA Center, University of Utah
Locations (15):
- United States (5):
  - Florida Heart Rhythm Institute, Tampa, Florida
  - Loyola University Medical Center, Chicago, Illinois
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute (Centennial), Nashville, Tennessee
- Royal Adelaide Hospital, Norwood, South Australia, Australia
- Universitair Ziekenhuis Ghent, Ghent, Belgium
- Hôpital Cardiologique du Haut-Lévêque/Bordeaux, Bordeaux, France
- Germany (5):
  - Kerckhoff Klinik, Bad Nauheim
  - Coburg Klinik, Coburg
  - Institut für Diagnostische und Interventionelle Radiologie - koln, Cologne
  - Asklepios Klinik St. Georg, Hamburg
  - Universitatsklinikum Leipzig, Leipzig
- St Antonius Ziekenhuis Hospital, Nieuwegein, Netherlands
- Hospital Clinic de Barcelona, Barcelona, Catalonia, Spain

REFERENCES:
- [Background] Oakes RS, Badger TJ, Kholmovski EG, Akoum N, Burgon NS, Fish EN, Blauer JJ, Rao SN, DiBella EV, Segerson NM, Daccarett M, Windfelder J, McGann CJ, Parker D, MacLeod RS, Marrouche NF. Detection and quantification of left atrial structural remodeling with delayed-enhancement magnetic resonance imaging in patients with atrial fibrillation. Circulation. 2009 Apr 7;119(13):1758-67. doi: 10.1161/CIRCULATIONAHA.108.811877. Epub 2009 Mar 23. PMID 19307477
- [Background] McGann CJ, Kholmovski EG, Oakes RS, Blauer JJ, Daccarett M, Segerson N, Airey KJ, Akoum N, Fish E, Badger TJ, DiBella EV, Parker D, MacLeod RS, Marrouche NF. New magnetic resonance imaging-based method for defining the extent of left atrial wall injury after the ablation of atrial fibrillation. J Am Coll Cardiol. 2008 Oct 7;52(15):1263-71. doi: 10.1016/j.jacc.2008.05.062. PMID 18926331
- [Background] Segerson NM, Daccarett M, Badger TJ, Shabaan A, Akoum N, Fish EN, Rao S, Burgon NS, Adjei-Poku Y, Kholmovski E, Vijayakumar S, DiBella EV, MacLeod RS, Marrouche NF. Magnetic resonance imaging-confirmed ablative debulking of the left atrial posterior wall and septum for treatment of persistent atrial fibrillation: rationale and initial experience. J Cardiovasc Electrophysiol. 2010 Feb;21(2):126-32. doi: 10.1111/j.1540-8167.2009.01611.x. Epub 2009 Oct 5. PMID 19804549
- [Background] Calkins H, Brugada J, Packer DL, Cappato R, Chen SA, Crijns HJ, Damiano RJ Jr, Davies DW, Haines DE, Haissaguerre M, Iesaka Y, Jackman W, Jais P, Kottkamp H, Kuck KH, Lindsay BD, Marchlinski FE, McCarthy PM, Mont JL, Morady F, Nademanee K, Natale A, Pappone C, Prystowsky E, Raviele A, Ruskin JN, Shemin RJ; Heart Rhythm Society; European Heart Rhythm Association; European Cardiac Arrhythmia Society; American College of Cardiology; American Heart Association; Society of Thoracic Surgeons. HRS/EHRA/ECAS expert consensus statement on catheter and surgical ablation of atrial fibrillation: recommendations for personnel, policy, procedures and follow-up. A report of the Heart Rhythm Society (HRS) Task Force on Catheter and Surgical Ablation of Atrial Fibrillation developed in partnership with the European Heart Rhythm Association (EHRA) and the European Cardiac Arrhythmia Society (ECAS); in collaboration with the American College of Cardiology (ACC), American Heart Association (AHA), and the Society of Thoracic Surgeons (STS). Endorsed and approved by the governing bodies of the American College of Cardiology, the American Heart Association, the European Cardiac Arrhythmia Society, the European Heart Rhythm Association, the Society of Thoracic Surgeons, and the Heart Rhythm Society. Europace. 2007 Jun;9(6):335-79. doi: 10.1093/europace/eum120. No abstract available. PMID 17599941